CLINICAL TRIAL: NCT05982288
Title: The Effect of Virtual Reality Software on Intensive Care Patient Care Management
Brief Title: Investigation of the Effect of Virtual Reality Software on Nurses' Clinical Practice, Problem Solving and Clinical Decision Making Skills and Anxiety in the Care Management of Intensive Care Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Banu Terzi, Associate Professor, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VR_BANUTERZI07
Record Dates: First submitted 2023-07-08; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Nurse's Role; Anxiety; Nursing Caries
Keywords: Problem solving; Clinical decision making; Intensive care nurses; Patient comfort; Critical decision making; Anxiety; Virtual reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a single-center, randomized controlled experimental design.
Masking Description: In this study, the single-blind method will be used to prevent nurses from interacting with each other. For this, the interventions will be performed on the same day and time using different areas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive care nurses (Experimental): Type of Study: It will be conducted in a single-center, randomized controlled experimental design. A clinical trial number will be obtained before starting the study.
  Location of the Study: The research will be conducted in the Anesthesiology and Reanimation Clinic of Antalya Kepez State Hospital.
  Interventions: Other: Virtual Reality Software

INTERVENTIONS:
Other: Virtual Reality Software — Training of intensive care nurses with virtual reality software

SUMMARY:
In the light of technological developments, learner-centered methods have begun to replace traditional teaching methods. Simulation applications are increasing in order to ensure patient safety and improve the quality of care in the training of nurses. Virtual reality, which is one of the simulation applications, is defined as an interactive, fun and virtual environment with three-dimensional visual feedback consisting of different sensory stimuli, where computer software and hardware are used together. When the studies on virtual reality, which is seen as a treatment, care and education tool in health care services, are examined; It is seen that virtual reality is mostly used in the teaching of some basic skills and in the education of nursing/medical students. From this point of view, in this project, which was submitted to the proposal, it was aimed to develop a virtual reality software for the care management of the intensive care patient and to investigate the effect of this software on the new intensive care nurses. Nurses to be included in the study will be randomly assigned to the control (n=34) and study groups (n=34). The research will be carried out in the following steps: 1) According to Kolcaba's Comfort Theory, the patient case scenario including the care management of the intensive care patient will be prepared and transferred to the virtual reality software, 2) The nurses in both groups will be given theoretical training on the care management of the intensive care patients, 3) The nurses forming the control group will be given theoretical training. A routine orientation training program will be given, and virtual reality glasses will be applied to the study group 4) "Knowledge Level Questionnaire", "Clinical Practice Skill Observation Form", "Problem Solving" before the theoretical training, 1 week after the application and in the first month of the application for both groups. Inventory", "Clinical Decision Making Scale in Nursing", "State Anxiety Inventory" and "Satisfaction Level Questionnaire" will be applied. With the software planned to be developed within the scope of the project, it is predicted that patient comfort and quality of life in intensive care will increase by providing rapid orientation to the clinic of the new intensive care nurses and increasing their clinical practice, problem solving and clinical decision making skills.

DETAILED DESCRIPTION:
The importance of qualified nurses in providing intensive care services and ensuring comfort cannot be denied. In this context, intensive care nurses are seen as the most important member and backbone of the interdisciplinary team. The realization of nurses' roles and responsibilities in the care management of patients in line with the nursing process, in line with evidence-based practices and guidelines, reduces the possible complications that may develop due to hospitalization in the intensive care unit . The prerequisite for providing quality and safe care in intensive care is that 75% of intensive care unit staff should be composed of specially trained nurses . During the training of nurses working in intensive care units, which is a specialized field, today's changing technology should be kept up with. The most effective and efficient way to do this is to develop continuous education opportunities. However, in addition to the problems experienced in accessing continuing education opportunities due to reasons such as responsibilities related to work and family life, unsuitability of working hours and places, and workload, the fact that learning methods continue mostly with traditional methods can make the situation difficult.

Increasing knowledge in line with technological developments reveals the necessity of "learner-centered methods" beyond traditional teaching methods. Especially in recent years, there has been an increasing interest in simulation applications to improve patient safety and patient care in the education of health care providers/nurses. Simulation applications give students the opportunity to realize complex learning objectives, demonstrate their competencies and be objectively evaluated in a realistic clinical environment without harming the patient. At the same time, many factors such as the inadequacy of clinical practice areas and the number of learners require the inclusion of simulation applications in nursing education. It is emphasized that virtual reality applications, which are one of the simulation applications for the continuous and professional development of learners / nurses, who are called digital natives today, are taking their place in these programs and will increase gradually in the future. It is stated that health technologies will contribute to healthcare professionals making fewer mistakes, accelerating the healing process of patients, increasing the quality and efficiency of health services, and that virtual reality technology will have an important place among the important technologies and trends that will affect the field of health until 2025. It is defined virtual reality as a virtual environment consisting of different sensory stimuli by combining computer software and hardware, while virtual reality used in healthcare is defined as a treatment, care and education tool with interactive, fun and three-dimensional visual feedback. The area of use of virtual reality application, which first started to be applied with video games, is gradually expanding. Since the most important feature that distinguishes virtual reality from other learning methods is that it gives a real feeling in practice, it acts as a bridge between theory and practice in nursing education. Virtual reality, which is not expensive to implement and use in education, does not cause side effects, is non-invasive, and has an effective role in physical, psychological, social, emotional and spiritual recovery, is not a choice but a necessity in current and future nursing practices and education.

In the light of all this information, it is important that intensive care nursing is a specialized field / branch, post-graduate education should be certified, critical thinking skills should be developed, critical patients' care needs should be met, and continuous training should be supported in order to adapt to changing and developing technology, care and treatment methods. The World Federation of Intensive Care Nurses Associations and the European Federation of Intensive Care Nurses Associations recommend that the care of the intensive care patient should be carried out by nurses specialized in intensive care nursing with postgraduate programs. It is known that a qualified intensive care nurse should receive at least 1200 hours of training after graduation and is trained in an average of five years. The intensive care nursing certificate program standards prepared in line with the Ministry of Health's Regulation on Certified Education aim to "train intensive care nurses who ensure the physical, psychological and social empowerment of the individual with preventive, developmental / rehabilitative interventions, establish therapeutic communication with patients and their families, adapt to developments in health science and technology, new treatment and care methods, have competence to meet emergency, critical and complex patient care needs, and have advanced problem-solving skills". In the training program, it is listed that learning methods such as oral lecture, video teaching, small group work, demonstration, active discussion with question-answer, simulation and clinical practice can be used.

Orientation programs have an important place in the adaptation process of newly graduated nurses to their professional roles. Orientation training consists of a comprehensive and intensive program that is based on the learning needs of newly graduated nurses, meets their expectations from the institution/profession, facilitates their adaptation to the profession/unit, provides competence to novices, and increases institutional commitment and job satisfaction. In orientation training, the scope, content and duration of which vary from institution to institution and according to the unit worked in, it is stated that the orientation period varies between 6 weeks and 12 months; in specialized units such as emergency, intensive care, etc., this period can increase from 12 weeks to 18 months.

Intensive care nurses have the opportunity to improve their competencies in basic knowledge and practice skills with clinical orientation training, competencies in advanced knowledge and practice skills with in-service training, and professionalism with certificates and courses. It is seen that most of the studies conducted abroad on the education of intensive care nurses are related to the implementation and evaluation of orientation programs. Studies show that special orientation models focusing on critical thinking skills, patient care management and the development of self-esteem are utilized in the orientation training of intensive care nurses. In researches' country, research on continuing education activities for the training and development of intensive care nurses is limited. In these limited studies, although participation in trainings, especially in-service trainings, is considered partially sufficient, it is also noteworthy that they cannot participate in trainings due to workload and lack of staff. In addition to these findings, the fact that the majority of the training method is lecture with slides is an indication that today's education system is based on traditional knowledge and this is reflected in continuing education activities such as orientation training and in-service training.

Studies show that the stress levels of newly graduated nurses whose first working experience is in specialized units such as intensive care, emergency, etc. are higher. However, when the literature is examined, it is seen that a significant portion of newly graduated nurses are directly assigned to specialized units. In the a study, 11% of newly graduated nurses worked in intensive care and 16% in emergency services; in the an other study, 16% worked in intensive care and 9% in emergency services; and in the other study, it was reported that 77% of newly graduated nurses were first assigned to specialized units such as intensive care, emergency, oncology, etc. Considering that newly graduated nurses start their professional practice with basic level professional knowledge and skills, specialized units such as intensive care, emergency service and oncology put more pressure on new graduates. This situation causes newly graduated nurses to feel professionally inadequate, experience intense stress and leave the profession/institution in the future. In researches' country, as in the international arena, it is seen that newly graduated nurses mostly start working in specialized units such as intensive care, emergency, etc. . In another study, it was determined that the area where new graduate nurses felt least competent was intensive care units and that they needed training specific to this area.

In the literature, there are studies in which virtual reality method is used in nursing education, and it is seen that these studies are mainly aimed at nurse students.

Virtual reality applications enable participants to learn interactively and analyze problems by increasing the learning outcomes for all learning areas (cognitive, affective, psychomotor) in educational institutions, increasing the permanence of learning. As seen in other studies, it is thought that the use of virtual reality in trainings organized for intensive care nurses in health institutions can increase the quality of care, increase patient comfort, reduce the error rate, reduce the stress level of learners and provide psychomotor skills. In addition, virtual reality applications can be used as a unique and useful alternative teaching method for intensive care nurses to gain more advanced and abstract skills such as collaboration, problem solving, critical thinking or communication skills and to evaluate these skills.

ELIGIBILITY:
Inclusion Criteria:

* To be a new graduate from the Department of Nursing
* Being a new employee in the intensive care unit
* Not having worked in an intensive care unit before
* Being willing and volunteering to participate in the study

Exclusion Criteria:

* Having just started working in the intensive care unit and subsequently changed duty station
* Resignation at any stage of the study
* Being a member of a profession other than nursing (midwife, ATT, paramedic, etc.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical practice skills questionnaire | 1-8 month
  Change in clinical practice skills of intensive care nurses
Problem-solving skills scale | 1-8 month
  The problem solving inventory is a scale consisting of a total of 35 items with 6 subgroups. The subgroups are as follows: hasty approach, thinking approach, avoidant approach, evaluative approach, self-confident approach and planned approach. Each group can be used independently. High total scores obtained from the whole scale indicate that the individual perceives himself/herself as inadequate in problem solving skills. The marking of the PSI is done on a 6 Likert-type scale. 21 items are scored as straight and 14 items are scored as reversed. The minimum score for the whole scale is 32 and the maximum score is 192. Items 9, 22 and 29 are excluded during scoring. Cronbach's alpha values found in the existing studies on the reliability of the scale are between 0.73 and 0.94.
The clinical decision making scale in nursing | 1-8 month
  The Clinical Decision Making Scale in Nursing consists of 40 items and four subscales. The subscales of the scale are "Exploring options and ideas", "Investigating goals and values", "Evaluating outcomes", and "Searching for information and adopting new information impartially". Each subscale consists of 10 items. The total scale is scored between 40 and 200 and each subscale is scored between 10 and 50 and there is no cut-off point. A high score on the scale indicates a high perception of decision making and a low score indicates a low perception of decision making. The evaluation of the scale is based on each subscale and the total score of the scale.
State anxiety scale | 1-8 month
  State Anxiety Scale is the subjective fear that an individual feels due to the stressful (pressurized) situation in which he/she is in. This scale can be applied to individuals over the age of 14. The inventory has two separate scales of 20 items each. State Anxiety Scale; determines how the individual feels at a certain moment and under certain conditions. It can be applied individually and as a group. In answering the State Anxiety Scale, it is asked to choose one of the options "not at all", "a little", "a lot" and "completely" according to the severity of the feelings, thoughts or behaviors expressed by the items. The total score value obtained from the scale varies between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Satisfaction questionnaire | 1-8 month
  In order to evaluate the satisfaction of the nurses with the virtual reality software, there are 10 items in the form prepared by the researchers in 3-point Likert type. The lowest and highest scores that can be obtained from the scale vary between 0-30. A total score of 15 above indicates a high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Terzi, PhD, Study Director — Akdeniz University
Locations (1):
- Kepez State Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
With the virtual reality software developed within the scope of the project, the effects of the training given to intensive care nurses in the care management of the intensive care patient on the clinical practice skills, problem solving skills, clinical decision making skills, anxiety levels and satisfaction levels of nurses will be examined.